CLINICAL TRIAL: NCT00862030
Title: Comparison of Two-versus Three-Dimensional Treatment Planning for Patients Receiving Chest Radiotherapy for Symptom Control
Brief Title: CT-Based Versus Conventional Simulation for Palliative Radiotherapy of Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alberta Health services (Other)
Responsible Party: Dr.Alysa Fairchild, Alberta Cancer Board
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: 24639
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Palliative radiotherapy; Treatment planning; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Study Cohort
  Interventions: Procedure: CT- simulation scan

INTERVENTIONS:
Procedure: CT- simulation scan — Patients who are receiving standard palliative radiotherapy planned under x-rays will also undergo 1 CT-simulation scan which they would otherwise not require. The planning x-rays and CT scan will then be compared dosimetrically

SUMMARY:
Radiotherapy (RT) treatment to the chest is a standard way of trying to decrease symptoms like cough or shortness of breath. Before any RT can be delivered, it must be planned, either using conventional x-rays ("fluoroscopy") or using computer tomography ("CT") scanning. This study is being done because the investigators do not know which of these two common ways of RT planning is better for balancing both treating the cancer and decreasing side effects.

DETAILED DESCRIPTION:
Standard RT planning will be performed under conventional simulation, followed by CT-simulation (for study purposes only). Retrospectively, 3D treatment fields will be designed using the CT-simulation data, and compared to the actual treatment fields planned using x-rays. Coverage of the tumour volume will be assessed, together with doses, field sizes and beam positions, to determine relative undercoverage of tumour and overcoverage of normal tissue between the two planning methods, if any.

ELIGIBILITY:
Inclusion Criteria:

* Patients with local symptoms secondary to histologically-confirmed non-small cell lung cancer
* Patients who will be receiving palliative-intent external beam radiotherapy
* Patients who are clinically appropriate for conventional radiotherapy planning
* Patients who can provide written informed consent

Exclusion Criteria:

* Patients who cannot provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alysa Fairchild, MD FRCPC, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada